CLINICAL TRIAL: NCT04147806
Title: A Pilot Study of Ultra-High-Dose Hypofractionated or Single-Dose Radiotherapy for Intermediate Risk Prostate Cancer
Acronym: PROSINT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-6545
Record Dates: First submitted 2019-10-10; First posted 2019-11-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dexamethasone; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- IGRT 45 Gy in 5 fractions of 9 Gy (Active Comparator): Hypofractionated IGRT at a prescription dose of 45 Gy in 5 fractions of 9 Gy delivered in five consecutive days
  Interventions: Radiation: IGRT 45 Gy in 5 fractions of 9 Gy; Radiation: IGRT 24 Gy single dose; Drug: Dexamethasone; Drug: Tamsulosin
- IGRT 24 Gy single dose (Experimental): single fraction IGRT at a prescription dose of 24 Gy
  Interventions: Radiation: IGRT 45 Gy in 5 fractions of 9 Gy; Radiation: IGRT 24 Gy single dose; Drug: Dexamethasone; Drug: Tamsulosin

INTERVENTIONS:
Radiation: IGRT 45 Gy in 5 fractions of 9 Gy — Administration of 9 Gy in five consecutive days, to a total dose of 45 Gy radiation
Radiation: IGRT 24 Gy single dose — Administration of a single dose of 24 Gy in one session
Drug: Dexamethasone — 4 mg by mouth on treatment days only
  Other Names: Dexasone
Drug: Tamsulosin — 0.4 mg by mouth daily starting the day of simulation and until 2 weeks post-treatment.
  Other Names: Flomax Relief

SUMMARY:
The present study evaluates clinical outcomes and treatment-related toxicity following definitive ultra-high dose external beam radiotherapy delivered with two different regimens in patients with intermediate-risk adenocarcinoma of the prostate. Modern computer-driven technology enables the implementation of ultra-high hypofractionated Image-Guided Radiotherapy (IGRT) safely.

Prostate cancer patients classified according to the current National Comprehensive Cancer Network (NCCN) guidelines as intermediate risk (biopsy Gleason score of 7 and/or Prostate Specific Antigen (PSA) level >10 and ≤20 ng/mL and/or Stage T1, T2a, T2b or T2c) are eligible for this study.

Patients will undergo IGRT with volumetric intensity-modulated arc radiotherapy (VMAT) with state-of-the-art treatment-planning and quality assurance procedures. Emphasis is placed on normal tissue sparing and delivery accuracy via the use of devices that ensure stability and beam location reproducibility. A rectal balloon with air filling will be used for prostate target immobilization and anatomical reproducibility, while a urethral catheter loaded with beacon transponders will be used to ensure set-up reproducibility and online target tracking. Previously untreated patients with intermediate-risk prostate cancer will be prospectively randomized to receive either 45 Gy in five fractions of 9 Gy each vs. 24 Gy in a single-dose.

Patients will be followed at one month post-treatment and every 3 months for up to 12 months (+/- 4 weeks) and every 6 months thereafter. Acute and chronic toxicity evaluations will focus on urinary, rectal and sexual functions and will be assessed through validated questionnaires. Serum PSA values will be regularly acquired during follow-up. A multiparametric MRI will be performed at baseline, 6, 12 and 24 months following intervention. Additionally, a post-treatment diffusion-weighted MRI (DW-MRI) will be performed within 15 minutes of the first treatment, to measure early physiologic changes, such as perfusion and ischemia, that may correlate with clinically relevant end-points. Post-treatment prostate needle biopsies will be obtained at 24 months to evaluate pathologic response to therapy. The study will be continuously monitored for a minimum of 5 years. In the event unexpected severe (grade ≥3) toxicities are observed in any one of the treatment arms, the study will be terminated according to the stopping rule >3/first 15 patients.

DETAILED DESCRIPTION:
This is open label feasibility study where patients enrolled in the study will undergo image-guided, intensity-modulated radiotherapy using the same equipment, techniques, and treatment-planning procedures as currently practiced at CCU. Eligible patients will receive either 45 Gy in 5 sessions each of 9 Gy delivered in one week (arm A) or 24 Gy in 1 session (arm B) to assess the dose limiting toxicities in the two groups. Patients will be randomized to arm A or arm B.

Dose limiting toxicity (DLT) is defined as any Grade 3 urinary or rectal toxicity, based on NCI CTCAE v4.0, observed within 3 months of completion of protocol radiation. If, at any point in the conduct of the trial, DLTs are observed in three patients in a study arm, accrual to that arm will be terminated.

There are three aspects of this study that will be different from the currently used standard treatment for definitive external beam treatment of prostate cancer:

1. The dose-fractionation scheme, as per the treatment arm.
2. Acquisition of a set of prostate biopsies at 24 months post treatment
3. Examination of imaging response based on multi-parametric MRI

ELIGIBILITY:
Inclusion Criteria:

* Signed study specific informed consent form;
* Histologic confirmation of adenocarcinoma of the prostate by biopsy;
* PSA ≤ 20 ng/mL;
* Gleason score 7;
* Staging MRI must confirm American Joint Committee on Cancer (AJCC) stage T1, T2a, T2b or T2c;
* No direct evidence of regional or distant metastases after appropriate staging studies;
* Age ≥ 50;
* Performance Status 0-2;
* Internation Prostate Symptom Score score must be ≤ 15 (alpha blockers allowed);
* CT scan or Ultrasound-based volume estimation of prostate gland ≤ 100 grams;

Exclusion Criteria:

* Positive lymph-nodes or metastatic disease from prostate cancer on imaging studies
* Prior invasive malignancy unless disease-free for a minimum of 5 years
* Tumour Clinical stage T3 or T4 on MRI
* PSA > 20 ng/mL
* Gleason score > 7
* Previous pelvic radiotherapy
* Previous surgery for prostate cancer
* Previous transurethral resection of the prostate (TURP)
* History of Crohn's Disease or Ulcerative Colitis
* Previous significant urinary obstructive symptoms
* Significant psychiatric illness
* Ultrasound or CT estimate of prostate volume > 100 grams
* Severe, active co-morbidity

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2026-07-13 (Estimated); Study Completion 2026-07-13 (Estimated)

PRIMARY OUTCOMES:
Number of patients with treatment-related adverse events as assessed by Common Toxicity Criteria for Adverse Effects v4.0 | Participants should be followed continuously, for the duration of 5 years
  Comparison of treatment related adverse events as measured by Common Toxicity Criteria for Adverse Effects v4.0 over a 5 year time frame

SECONDARY OUTCOMES:
Biochemical outcome based on Prostate Specific Antigen (PSA) assessment | Participants should be followed continuously for the duration of 5 years
  PSA assessment will be done
Quality of life assessment based on International Prostate Symptom Score (IPSS) | Participants should be followed continuously for the duration of 5 years
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms.The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Pathological response based on biopsy at 24 months post-treatment | Participants should be followed continuously for the duration of 5 years
  Pathology will be evaluated
Quality of life assessment based on International Index of Erectile Function (IIEF) | Participants should be followed continuously for the duration of 5 years
  Quality of life survey

CONTACTS AND LOCATIONS:
Overall Officials: Madhur Garg, MD, Principal Investigator — Associate Clinical Director
Locations (1):
- Montefiore Medical Center - Moses Campus, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No